CLINICAL TRIAL: NCT03914027
Title: Feasibility & Effect of a Tele-rehabilitation Program in Pulmonary Sarcoidosis
Brief Title: Feasibility & Effect of a Tele-rehabilitation Program in Pulmonary Sarcoidosis Pulmonary Sarcoidosis
Acronym: TeleSarco
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: Eurostars (Other); University of Aarhus (Other)
Responsible Party: Principal Investigator, Jose Cerdan, PhD student, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TeleSarco
Record Dates: First submitted 2019-04-08; First posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Sarcoidosis, Pulmonary; Telerehabilitation
MeSH Terms: conditions — Sarcoidosis, Pulmonary | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial. 24 patients with PS will be randomized in two groups, trained by tele-rehabilitation for 12 weeks and afterwards followed for 6 months. The control group will follow the usual control program for PS patients that only involves outpatient visits approximately every 3rd month. No specific PS rehabilitation program exists. The intervention group will receive TR in the form of video consultations- and chat sessions with a real physiotherapist and workout sessions with a virtual physiotherapist agent. They will also train with virtual reality glasses or tablets that show the actual exercises in the training program.
Who Masked: Participant, Investigator
Masking Description: Randomisation will allocate patients to either the intervention or control group. This will be performed electronically by using a randomization plan generator ("Randomization Plans: Never the Same Thing Twice!" n.d.) that has already given a randomization plan and code to generate the same plan obtained. To reproduce this study randomization plan, enter at http://www.jerrydallal.com/random/permute.htm :
  24 subjects randomized into 2 blocks (intervention, control) Seed number 10180. Block randomization will be used to ensure that the numbers of participants assigned to each group is equally distributed during the different seasons.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Patients allocated to the control group will follow the same procedure except for not using tele-rehabilitation.
- Intervention (Experimental): The intervention is the use of a tele-rehabilitation program during 12 weeks. The patient's training time will be registered automatically. The control group will receive standard treatment only.
  Interventions: Behavioral: Telerehabilitation

INTERVENTIONS:
Behavioral: Telerehabilitation — Each patient will have the opportunity to have minimum one VC per week the first month, one Video Consultation each second week the second month one VC a month the rest of the trial. Here the physiotherapist, via history will extract the information needed to calibrate the daily TR program according to the patient's physical status and needs.
  Workout Sessions with a Virtual Physiotherapist Agent (VPA): The patient will train according to what is decided by the physiotherapist and the patient in the VC or chat meetings. Normally, the patients will train 10-20 minutes daily at home with its individual and tailored VPA. Instead of ergometer bike training, the patient will receive some easy training tools such as elastics, weights and a fitness-step that can be used in the different exercises showed by the VPA to reach the same intensity of workout. The VPA will then be animated to motivate and encourage the patient to exercises at home.
  Other Names: remote rehabilitation
  Arms: Intervention

SUMMARY:
Pulmonary sarcoidosis (PS) is defined as a multisystem granulomatous disorder of unknown cause affecting different vital organs, especially the lungs.

PS manifest in reduction of pulmonary function. Overall symptoms lead to poor physical conditioning contributing to a vicious cycle of more physical inactivity.

Treatment of sarcoidosis is usually limited to patient symptoms. Progressive fibrosis sometimes can lead to respiratory failure and ultimately, pulmonary transplantation.

Physical training shows promising evidence of a positive effect on PF. No defined training program with regard to exercise frequency, duration or intensities exists.

PS is a relatively rare disease and patients are scattered in great geographically areas,.It is difficult to organize targeted group training with supervised physical training, convenient for patients and affordable for the public health sector. Tele-rehabilitation (TR) seems to be a good approach to reach patients in low inhabited areas, going from health care to self-care, empowering patient's awareness of their disease and increasing the flexibility patients need to acquire healthier behaviors.

Preliminary evaluations from TR initiatives in Scotland showed tele-rehabilitation to be more cost effective with patients living in remote areas than with the outreach- or centralized model.

No studies on the feasibility effect of TR in PS exists. The study is a prospective randomized controlled trial investigating the effects of tele-rehabilitation in patients with PS compared to standard practice. 24 patients with PS will be randomized in two groups, trained by tele-rehabilitation for 12 weeks and afterwards followed for 6 months. The control group will follow the usual control program for PS patients that only involves outpatient visits approximately every 3rd month. No specific PS rehabilitation program exists. The intervention group will receive TR in the form of video consultations- and chat sessions with a real physiotherapist and workout sessions with a virtual physiotherapist agent. They will also train with virtual reality glasses or tablets that show the actual exercises in the training program.

Patients will be tested with pulmonary function, physical, anxiety and quality of life parameters, all at baseline, after 12 weeks of intervention, 3 and 6 months after cessation of the program.

DETAILED DESCRIPTION:
Background:

Pulmonary Sarcoidosis (PS) is defined as a multisystem granulomatous disorder of unknown cause affecting different vital organs, especially the lungs . The pathogenesis is complex and a single immunologic reaction and modulation of one cytokine is unlikely to resolve all aspects of the disease.

PS affects people throughout the world. The prevalence in Denmark is 6.4 cases per 100,000, consistent with the range of 5 to 40 per 100,000 reported from other northern European countries.

PS manifest in reduction of pulmonary function resulting in cough, dyspnea and fatigue and can be complicated by fibrosis and pulmonary hypertension. The overall symptoms lead to poor physical conditioning contributing to a vicious cycle of more physical inactivity

Treatment of sarcoidosis is usually limited to patient symptoms. In case of progressive pulmonary involvement or involvement of other vital organs, corticosteroids are indicated to prevent or stabilize organ damage. However, progressive fibrosis sometimes can lead to respiratory failure and ultimately, pulmonary transplantation.

Physical training shows promising evidence of a positive effect on PF, can improve psychological health and physical functioning and also decrease fatigue, increase muscle strength and increase exercise capacity. Until today there is no defined training program with regard to exercise frequency, duration or intensities in PS contrary to chronic obstructive pulmonary diseases (COPD) or idiopathic pulmonary fibrosis (IPF).

PS is a relatively rare disease and that sarcoid patients are scattered in great geographically areas, it is difficult to organize targeted group training with supervised physical training, convenient for patients and affordable for the public health sector. New technologies in healthcare are being introduced to treat patients from a distance in these years. Tele-rehabilitation (TR) seems to be a good approach to reach patients in low inhabited areas, going from health care to self-care, empowering patient's awareness of their disease and increasing the flexibility patients need to acquire healthier behaviors. TR has previously been shown to be feasible in patients with lymphedema, COPD and orthopedic diseases for lower back, knee and shoulder.

TR with COPD patients at home is feasible and well accepted by the patients, although technology has been perceived as difficult. TR seems to improve the functional level as assessed by walking capacity, dyspnea, quality of life and daily physical activity . The interaction between the COPD patients at home and the healthcare professionals at the clinic through TR has evolved as a dialogue channel forming a basis for mutual learning processes and new relationships. Preliminary evaluations from TR initiatives in Scotland showed tele-rehabilitation to be more cost effective with patients living in remote areas than with the outreach- or centralized model.

There have so far been no studies on the feasibility effect of TR in PS.

Hypothesis Tele-rehabilitation in patients with PS is feasible and improves exercise capacity, quality of life and activities of daily living.

Aim To assess the feasibility and effect of tele-rehabilitation with a tele-rehabilitation platform (NITRP) compared to standard treatment with respect to exercise capacity, quality of life and activities of daily living in patients with PS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PS
* Signed informed consent
* Adults ≥ 18 years
* DLCO ≥ 30% predicted and FVC ≥ 50% predicted
* 6 minute walking test distance ≥ 150 m

Exclusion Criteria:

* Participation in an official rehabilitation program < 3 months before start of the study Musculoskeletal disorders
* Severe cardiac diseases (ejection fraction < 30%, daily angina, or otherwise specified by treating cardiologist)
* Unable to understand informed consent
* Other conditions that hamper the use of tele-rehabilitation
* Non-Danish speaking.
* Unwillingness to implement the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
6MWT -12 weeks | 12 weeks afte baseline
  Change in the distance walked at a 6MWT measured at week 12.

SECONDARY OUTCOMES:
6MWT 6 and 9 month | 6 and 9 months after baseline.
  Change in the distance walked at a 6MWT 6 and 9 months after baseline.
Change in muscle strength measured with the MVC | 12 weeks, 6 and 9 months after baseline
  Change in muscle strength measured with the MVC of the dominant arm
Change in total score in health-related quality of life measured by Sct. Georges Respiratory Questionnaire (Jones, Quirk, and Baveystock 1991) (SGRQ) | 12 weeks, 6 and 9 months after baseline
  SGRQ is a disease specific, self-administered questionnaire with 50 items comprising two domains with 3 components as symptoms, activity and impacts. Each is scored from 0-100, with higher scores corresponding to worse health related quality of life.
Change in fatigue measured by 10-item Fatigue Assessment Scale (FAS) | 12 weeks, 6 and 9 months after baseline
  Change in fatigue measured by FAS at 12 weeks, 6 and 9 months after baseline. The 10-item Fatigue Assessment Scale (FAS)(Vries et al. 2004) (Michielsen et al. 2006) is a 10-item general fatigue questionnaire to assess fatigue. Five questions reflect physical fatigue and 5 questions (questions 3 and 6-9) mental fatigue. An answer to every question has to be given, even if the person does not have any complaints at the moment. Scores on question 4 and 10 should be recoded (1=5, 2=4, 3=3, 4=2, 5=1). Subsequently, the total FAS score can be calculated by summing the scores on all questions (recoded scores for questions 4 and 10). The total score ranges from 10 to 50. A total FAS score < 22 indicates no fatigue, a score ≥ 22 indicates fatigue. All online versions of the FAS calculate the FAS scores automatically: a total score as well as mental and physical score will be provided.
Change in total score in health-related quality of life measured by The King's Brief Interstitial Lung disease health status questionnaire (KBILD) | 12 weeks, 6 and 9 months after baseline
  Change in total score in health-related quality of life measured by KBILD at 12 weeks, 6 and 9 months after baseline
  The King's Brief Interstitial Lung disease health status questionnaire (Taylor et al. 2015) is a disease specific, validated, self-completed health status questionnaire that is comprised of 15 items. It has three domains: psychological, breathlessness, activities and chest symptoms. The KBILD domain and total score ranges are 0-100; 100 = best.
Change in total score of anxiety measured by The General Anxiety Disorder Score (GAD-7 ) | 12 weeks, 6 and 9 months after baseline
  Change in total score of anxiety measured by GAD-7 at 12 weeks, 6 and 9 months after baseline The General Anxiety Disorder Score (Jones, Quirk, and Baveystock 1991; Löwe et al. 2008) measures the presence and severity of general anxiety disorder. It is a 7 self-rated items, each item scores 0-3 (not at all, several days, more than half the days, nearly every day); total score range 0-21.
Change in component scores (symptoms, activity & impact) in health-related quality of life measured by SGRQ | 12 weeks, 6 and 9 months after baseline
  Change in component scores (symptoms, activity & impact) in health-related quality of life measured by SGRQ at 12 weeks, 6 and 9 months after baseline.
  The King's Brief Interstitial Lung disease health status questionnaire (Taylor et al. 2015) is a disease specific, validated, self-completed health status questionnaire that is comprised of 15 items. It has three domains: psychological, breathlessness, activities and chest symptoms. The KBILD domain and total score ranges are 0-100; 100 = best.
Change in the number of steps walked measured by a pedometer. | 12 weeks, 6 and 9 months after baseline
  Change in the number of steps walked measured by a pedometer.
Cost of the tele-rehabilitation program | 12 weeks after baseline
  Cost of the tele-rehabilitation program

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Bendstrup, PhD, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Pulmonary Disease Research Center, Aarhus, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633